CLINICAL TRIAL: NCT00410163
Title: An Open-labeled, Randomized, Two-dose, Parallel Group Trial of Ofatumumab, a Fully Human Monoclonal Anti-CD20 Antibody, in Combination With Fludarabine and Cyclophosphamide, in Patients With Previously Untreated B-cell CLL
Brief Title: Ofatumumab With Fludarabine and Cyclophosphamide in B-CLL Patients
Acronym: BIFROST
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 111774; Hx-CD20-407 (Other: Genmab); The BIFROST trial
Record Dates: First submitted 2006-12-11; First posted 2006-12-12 (Estimated); Results first posted 2011-10-17 (Estimated); Last update posted 2014-02-10 (Estimated); Status verified 2013-11

CONDITIONS: Leukaemia, Lymphocytic, Chronic
Keywords: B-cell; cyclophosphamide; fludarabine; Chronic Lymphocytic Leukemia; Ofatumumab
MeSH Terms: conditions — Leukemia, B-Cell; Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab; fludarabine; Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Active Comparator 1 (Active Comparator): Each patient will receive a total of 6 infusions with ofatumumab every 4 weeks in combination with fludarabine and cyclophosphamide. The first infusion will be 300mg followed by 5 infusions of 500mg
  Interventions: Drug: Ofatumumab 500mg; Drug: Fludarabine; Drug: Cyclophosphamide
- Active Comparator 2 (Active Comparator): Each patient will receive a total of 6 monthly infusions with ofatumumab in combination with fludarabine and cyclophosphamide. The first infusion will be 300mg followed by 5 infusions of 1000mg
  Interventions: Drug: Ofatumumab 1000mg; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Drug: Ofatumumab 500mg — Ofatumumab 500mg or should be diluted into 1000mL pyrogenefree saline and administered as an IV infusion.Duration of infusion will be approximately 6½ hours.Infusions should be given every 4 weeks until a total of 6 infusions has been given.
  Arms: Active Comparator 1
Drug: Ofatumumab 1000mg — Ofatumumab 1000mg or should be diluted into 1000mL pyrogenefree saline and administered as an IV infusion.Duration of infusion will be approximately 6½ hours.Infusions should be given every 4 weeks until a total of 6 infusions has been given.
  Arms: Active Comparator 2
Drug: Fludarabine — Fludarabine (25 mg/m2) should be administered as an IV infusion daily, Days 2 through 4 of Course 1, and Days 1 through 3 of Courses 2 through 6, every 4 weeks for 6 courses
Drug: Cyclophosphamide — Cyclophosphamide (250 mg/m2) should be administered as an IV infusion daily, Days 2 through 4 of Course 1, and Days 1 through 3 of Courses 2 through 6, every 4 weeks for 6 courses.

SUMMARY:
To investigate the safety and efficacy of two dose regimes of ofatumumab in combination with chemotherapy in previously untreated patients with B-CLL

ELIGIBILITY:
Inclusion Criteria:

1. Patients with active B-CLL and with an indication for treatment
2. Age ≥ 18 years
3. Following receipt of verbal and written information about the study, the patient must provide signed informed consent before any study related activity is carried out

Exclusion Criteria:

1. Any previous treatment for B-CLL or any other treatments that can be considered active against B-CLL
2. Glucocorticoid unless given in doses ≤ 10 mg /day for other indications than B-CLL (e.g. asthma)
3. Known transformation of B-CLL
4. Known CNS involvement of B-CLL
5. Past or current malignancy, except for:

   1. Cervical carcinoma Stage 1B or less
   2. Non-invasive basal cell and squamous cell skin carcinoma
   3. Malignant melanoma with a complete response of a duration of > 10 years
   4. Other cancer diagnoses with a complete response of a duration of > 5 years
6. Chronic or current infectious disease requiring systemic treatment
7. Clinically significant cardiac disease
8. Significant concurrent, uncontrolled medical condition
9. History of significant cerebrovascular disease
10. Known HIV positive
11. Positive serology for hepatitis B, unless due to vaccination
12. Leukapheresis, except as a safety measure before chemotherapy
13. ECOG Performance Status of 3 or 4
14. Patients who at the time of inclusion are not expected to be able to complete the ofatumumab-FC regimen
15. Patients who have received treatment with any non-marketed drug substance or experimental therapy within 4 weeks prior to Visit 1
16. Current participation in any other interventional clinical study
17. Patients known or suspected of not being able to comply with a study protocol (e.g. due to alcoholism, drug dependency or psychological disorder)
18. Breast feeding women or women with a positive pregnancy test at Visit 1
19. Women of childbearing potential not willing to use adequate contraception for up to one year after last dose of ofatumumab. Adequate contraception is defined as hormonal birth control or intrauterine device. For patients in the USA the use of a double barrier method is also considered adequate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2007-01; Primary Completion 2009-03 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- GSK Investigational Site, Houston, Texas, United States
- GSK Investigational Site, Plymouth, Devon, United Kingdom

REFERENCES:
- [Background] Wierda WG, Kipps TJ, Durig J, Griskevicius L, Stilgenbauer S, Mayer J, Smolej L, Hess G, Griniute R, Hernandez-Ilizaliturri FJ, Padmanabhan S, Gorczyca M, Chang CN, Chan G, Gupta I, Nielsen TG, Russell CA; 407 Study Investigators. Chemoimmunotherapy with O-FC in previously untreated patients with chronic lymphocytic leukemia. Blood. 2011 Jun 16;117(24):6450-8. doi: 10.1182/blood-2010-12-323980. Epub 2011 Apr 15. PMID 21498674
- [Background] Wierda WG, Kipps TJ, Dürig J, Griskevicius L, Stilgenbauer S, Mayer J et al.. Chemoimmunotherapy with Ofatumumab, Fludarabine and Cyclophosphamide (O-FC) in Previously Untreated Patients with Chronic Lymphocytic Leukemia (CLL). [Blood]. 2010;E pub ahead of print:
- [Derived] Jewell RC, Kipps TJ, Durig J, Griskevicius L, Stilgenbauer S, Smolej L, Mayer J, Hess G, Hernandez-Ilizaliturri FJ, Padmanabhan-Iyer S, Fang L, Goldstein N, Gorczyca M, Gupta I, Lisby S, Wierda WG; Hx-CD20-407 Study Investigators. Associations of ofatumumab exposure and treatment outcomes in patients with untreated CLL receiving chemoimmunotherapy. Leuk Lymphoma. 2017 Feb;58(2):348-356. doi: 10.1080/10428194.2016.1195497. Epub 2016 Jul 7. PMID 27389174

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants received up to 6 courses (22 weeks) of treatment. After treatment, participants were evaluated for up to 18 months in a follow-up (FU) period and then entered an extended FU phase (up to Month 60). The overall study period reported is from 09 January 2007 to 05 June 2013, when all phases of the study were completed.
Groups:
- Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC): Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg) for course 1, followed by dose of 500 mg for courses 2-6 in combination with fludarabine iv (25 mg/meters squared [m^2] daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses. After the last infusion, the disease status of the participants was evaluated every 3 months up to 18 months during the Follow-up Period. Participants were monitored in the Extended Follow-up Phase every 6 months for survival until alternative Chronic Lymphocyte Leukemia (CLL) therapy was initiated, or until Month 60.
- Ofatumumab 1000 mg + FC: Ofatumumab iv infusion initiated at 300 mg for course 1, followed by dose of 1000 mg for courses 2-6 in combination with fludarabine iv (25 mg/m^2 daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses. After the last infusion, the disease status of the participants was evaluated every 3 months up to 18 months during the Follow-up Period. Participants were monitored in the Extended Follow-up Phase every 6 months for survival until alternative CLL therapy was initiated, or until Month 60.
Period: Treatment and Follow-up Phase (2 Years)
Arm/Group | Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC) | Ofatumumab 1000 mg + FC
Started | 31 | 30
Completed | 19 | 19
Not Completed | 12 | 11
Not completed — Adverse Event | 4 | 2
Not completed — Death | 1 | 1
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Lack of Efficacy | 0 | 4
Not completed — Participant Had No Response | 2 | 1
Not completed — Participant Had Stable Disease | 1 | 0
Not completed — Participant Received New Therapy | 1 | 1
Not completed — Participant Had Bone Marrow Transplant | 1 | 0
Not completed — Investigator Decision | 0 | 1
Period: Extended Follow-up (FU) Phase (2-5 Years
Arm/Group | Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC) | Ofatumumab 1000 mg + FC
Started | 20 (Participants who withdrew from the Treatment Phase were eligible to enter the Extended FU Phase.) | 21 (Participants who withdrew from the Treatment Phase were eligible to enter the Extended FU Phase.)
Completed | 10 | 11
Not Completed | 10 | 10
Not completed — Lost to Follow-up | 3 | 1
Not completed — Death | 1 | 1
Not completed — Medical Reasons | 1 | 0
Not completed — New Anti-CLL Treatment | 4 | 8
Not completed — Secondary Acute Myeloid Leukemia | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Ofatumumab 500 mg + FC: Ofatumumab iv infusion initiated at 300 mg for course 1, followed by dose of 500 mg for courses 2-6 in combination with fludarabine iv (25 mg/m^2 daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses
- Ofatumumab 1000 mg + FC: Ofatumumab iv infusion initiated at 300 mg for course 1, followed by dose of 1000 mg for courses 2-6 in combination with fludarabine iv (25 mg/m^2 daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses
- Total: Total of all reporting groups
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC | Total
Number analyzed (Participants) | 31 | 30 | 61
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (8.4) | 56.4 (8.7) | 56.2 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 7 | 18
  Male | 20 | 23 | 43
Race/Ethnicity, Customized [Number; unit: participants]
  White | 31 | 29 | 60
  Black or African American | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (Par.) With Complete Remission (CR), Measured From Start of Treatment Until 3 Months After Last Infusion
Description: Par. were evaluated for response by an Independent Endpoint Review Committee (IRC) in accordance with the National Cancer Institute-sponsored Working Group (NCI-WG) 1996 guideline. Par. with Complete Remission (CR) were classified as "complete responders". As per NCI-WG, CR requires all of the following criteria for a period of >=2 months: absence of lymphadenopathy (all lymph nodes <1.0 centimeters), no hepatomegaly/splenomegaly, absence of constitutional symptoms, lymphocytes <=4.0*10^9/liter (L), neutrophil leukocytes >=1.5*10^9/L, platelets >100*10^9/L, and hemoglobin >11 grams/deciliter.
Time Frame: Start of treatment (Day 1 of Week 0) until 3 months after start of last infusion (up to Week 32)
Population: Full Analysis Set (FAS): all participants who had been exposed to study drug irrespective of their compliance to the planned course of treatment
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
participants | 10 | 15

2. Secondary Outcome: Duration of Response
Description: The duration of response was defined as the time from the initial response (the first visit at which response was observed) to progression or death. For participants who were lost to follow-up, duration of response was censored at the date of the last attended visit at which the endpoint was assessed.
Time Frame: From time of initial response to disease progression or death, whichever came first, assessed over 2 years
Population: FAS. Only those participants classified as responders were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ofatumumab 500 mg + FC: Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg) for course 1, followed by dose of 500 mg for courses 2-6 in combination with fludarabine iv (25 mg/meters squared [m^2] daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses
- Ofatumumab 1000 mg + FC: Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg) for course 1, followed by dose of 1000 mg for courses 2-6 in combination with fludarabine iv (25 mg/meters squared [m^2] daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 24 | 22
months | NA [NA to NA] — An insufficient number of participants experienced progression or death after response to reach a median or calculate a confidence interval. | NA [NA to NA] — An insufficient number of participants experienced progression or death after response to reach a median or calculate a confidence interval.

3. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival (PFS) was defined as the time from randomization until the first radiologically or clinically documented evidence of progression or death due to any cause, if sooner. For participants who were lost to follow-up, PFS was censored at the date of the last attended visit at which the endpoint was assessed. The Kaplan-Meier method was used to estimate PFS.
Time Frame: From time of randomization to first documented evidence of disease progression or death due to any cause, whichever came first, assessed over 2 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
months | NA [NA to NA] — An insufficient number of participants experienced progression or death to reach a median or calculate a confidence interval. | 23.5 [NA to NA] — An insufficient number of participants experienced progression or death to calculate a confidence interval.

4. Secondary Outcome: Time to Next Anti-chronic Lymphocytic Leukemia (CLL) Therapy or Death
Description: Time to next anti-CLL (anti-lymphoma) therapy was defined as the time from randomization until the time of first administration of the next anti-lymphoma therapy other than ofatumumab or death. For participants who were lost to follow-up, the time was censored at the date of the last attended visit at which the endpoint was assessed.
Time Frame: From time of randomization to first administration of next anti-CLL therapy other than ofatumumab or death, assessed over 5 years
Population: FAS
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
months | 33.4 [27.3 to 46.9] | 33.3 [26.7 to 54.6]

5. Secondary Outcome: Median Percent Change in Tumor Size From Baseline (Visit 2, Wk 0) at Visits 9, 21, 25, 29, 33, 34, 35, and 37
Description: Tumor size was measured by physical examination of palpable abnormal lymph nodes. Percent change from Baseline (Visit 2, Week 0) = (value at indicated visits minus value at Visit 2 divided by value at Visit 2) * 100. Visits 33, 34, 35, 36, and 37 are measured in the number of months from the start of the last infusion. The start of the last infusion could have occurred up to Week 20.
Time Frame: Baseline Visit 2 (Week [Wk] 0); Visits 9 (Wk 4), 21 (Wk 12), 25 (Wk 16), 29 (Wk 20), 33 (Month [M] 1 after start of last infusion [LI]), 34 (M 3 after start of LI), 35 (M 6 after start of LI), 36 (M 9 after start of LI), and 37 (M 12 after start of L
Population: FAS. Data were provided for the number of participants attending each visit. Participants withdrawn during the study were not analyzed.
Measure: Median (Full Range); unit: percent change in tumor size
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 29 | 28
percent change in tumor size
  Visit 9 (Week 4), n=29, 28 | -75.00 [-100.00 to 0.00] | -70.90 [-100.00 to 73.00]
  Visit 21 (Week 12), n=24, 23 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to -39.00]
  Visit 25 (Week 16), n=23, 20 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to -85.00]
  Visit 29 (Week 20), n=22, 16 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to -92.00]
  Visit 33 (Month 1), n=21, 24 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to -4.00]
  Visit 34 (Month 3), n=22, 23 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to -40.00]
  Visit 35 (Month 6), n=19, 22 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to 12.00]
  Visit 36 (Month 9), n=20, 22 | -100.00 [-100.00 to 0.00] | -100.00 [-100.00 to 28.00]
  Visit 37 (Month 12), n=20, 18 | -100.00 [-100.00 to -100.00] | -100.00 [-100.00 to -69.00]

6. Secondary Outcome: Median Percent Change in CD5+CD19+ and CD5+CD20+ Cells in Peripheral Blood From Onset of Course 3 Throughout Follow-up (FU) Compared to Screening
Description: Malignant B cells (CD5+CD19+ and CD5+CD20+) were measured in peripheral blood samples by flow cytometry. Percent change from Screening (Visit 1, Week -2) = (value at indicated visits minus value at Visit 1 divided by value at Visit 1) * 100. Visits 33 and 34 are measured in the number of months from the start of the last infusion. The start of the last infusion could have occurred up to Week 20.
Time Frame: Baseline Visit 2 (Week [Wk] 0); Visits 15 (Wk 8), 21 (Wk 12), 25 (Wk 16), 29 (Wk 20), 33 (Month [M] 1 after start of last infusion [LI]), 34 (M 3 after start of LI)
Population: as for outcome 5
Measure: Median (Full Range); unit: percent change in cells
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 25 | 26
percent change in cells
  CD5+CD19+ cells, Visit 15 (Wk 8), n=25, 26 | -100.00 [-100.0 to 22.0] | -100.00 [-100.00 to -81]
  CD5+CD19+ cells, Visit 21 (Wk 12), n=24, 24 | -100.00 [-100.00 to -84.00] | -100.00 [-100.00 to -90.00]
  CD5+CD19+ cells, Visit 25 (Wk16), n=23, 21 | -100.00 [-100.00 to -93.00] | -100.00 [-100.00 to -96]
  CD5+CD19+ cells, Visit 29 (Wk 20), n=22, 19 | -100.00 [-100.00 to -98] | -100.00 [-100.00 to -96]
  CD5+CD19+ cells, Visit 33 (Wk 24), n=21, 24 | -100.00 [-100.00 to -99.00] | -100.00 [-100.00 to -73]
  CD5+CD19+ cells, Visit 34 (Wk 32), n=20, 22 | -100.00 [-100.00 to -95] | -100.00 [-100.00 to -97]
  CD5+CD20+ cells, Visit 15 (Wk 8), n=25, 26 | -100.00 [-100.00 to 22.00] | -100.00 [-100.00 to -92]
  CD5+CD20+ cells, Visit 21 (Wk 12), n=24, 24 | -100.00 [-100.00 to -84] | -100.00 [-100.00 to -96]
  CD5+CD20+ cells, Visit 25 (Wk16), n=23, 21 | -100.00 [-100.00 to -93] | -100.00 [-100.00 to -100]
  CD5+CD20+ cells, Visit 29 (Wk 20), n=22, 19 | -100.00 [-100.00 to -99] | -100.00 [-100.00 to -100]
  CD5+CD20+ cells, Visit 33 (Wk 24), n=21, 24 | -100.00 [-100.00 to -99] | -100.00 [-100.00 to -97.00]
  CD5+CD20+ cells, Visit 34 (Wk 32), n=20, 22 | -100.00 [-100.00 to -96] | -100.00 [-100.00 to -97.0]

7. Secondary Outcome: Number of Participants Who Experienced Any Adverse Event From First Treatment (Visit 2) to Visit 43 (Month 60)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a participant administered a pharmaceutical product and which did not necessarily have a causal relationship with this treatment. A list of AEs experienced in the study at a frequency threshold of 5% can be found in the AE section.
Time Frame: From first treatment (Visit 2) up to Visit 43 (Month 60)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
participants | 31 | 30

8. Secondary Outcome: Number of Participants With Positive Human Anti-human Anti Bodies (HAHA) at Visits 1, 21, 35, and 39
Description: HAHA are indicators of immunogenicity to ofatumumab. Blood samples were drawn from participants at Visits 1, 21, 35, and 39 for analysis of HAHA. Analysis of HAHA was done in batches.
Time Frame: Visits 1 (Screening, Visit -2), 21 (Week 12), 35 (Month 6), and 39 (Month 18)
Population: as for outcome 5
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
participants
  Visit 1 (Week -2), n=31, 30 | 0 | 0
  Visit 21 (Week 12), n=24, 24 | 0 | 0
  Visit 35 (Month 6), n=19, 22 | 0 | 0
  Visit 39 (Month 18), n=14, 13 | 0 | 0

9. Secondary Outcome: Number of Participants Who Reported Myelosuppression (Anemia, Leukopenia, Neutropenia, and Thrombocytopenia)
Description: Myelosuppression is one of the expected AEs for FC treatment and is defined as the decrease in the ability of the bone marrow to produce blood cells. The number of participants with myelosuppression was assessed from laboratory measurements with Grades 3(severe)-4 (life-threatening/disabling) (1, mild; 2, moderate; 5, death) according to the Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0. The CTCAE is issued by the National Cancer Institute (NCI) and is the standard classification used for the severity grading scale for AEs in cancer therapy clinical studies.
Time Frame: From first treatment (Visit 2) up to Visit 43 (Month 60)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
participants
  Anemia | 6 | 8
  Leukopenia | 23 | 22
  Neutropenia | 29 | 26
  Thrombocytopenia | 4 | 8

10. Secondary Outcome: Percent Change From Screening (Visit 1) in Complement (CH50) Levels at Visit 9 (Week 4)
Description: Blood samples were drawn from participants at Visits 1 and 9 for analysis of complement (CH50) levels. Analysis of CH50 was done in batches, and CH50 levels were measured two hours after the end of study medication infusion. Percent change from Screening (Visit 1, Week -2) = (value at Visit 9 minus value at Visit 1 divided by value at Visit 1) * 100.
Time Frame: Visit 1 (Week -2) and Visit 9 (Week 4)
Population: FAS. Data were provided for the number of participants attending Visit 9. Participants withdrawn during the study were not analyzed.
Measure: Median (Full Range); unit: Percent change in complement levels
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 29 | 26
Percent change in complement levels | 0 [-54 to 520] | 0 [-83 to 430]

11. Primary Outcome: Number of Participants (Par.) Who Were Classified as Responders and Non-responders
Description: Par. were evaluated by an IRC in accordance with NCI-WG 1996 guideline. Responders: CR, Nodular Partial Remission (nPR, same as CR, but persistent bone marrow nodules), and Partial Remission (PR, >=50% decrease in lymphocytes from pretreatment baseline (BL) value, >=50% reduction in lymphadenopathy, >=50% reduction of liver/spleen and neutrophils >= 1.5*10^9/L or platelets >100*10^9/L or hemoglobin >11 g/dL (or 50% improvement over BL for neutrophils, platelets, hemoglobin); non-responders: Stable Disease (SD, did not achieve CR/PR, and no PD), Progressive Disease (PD), or Not Evaluable (NE).
Time Frame: From start of treatment (Day 1 of Week 0) until 3 months after start of last infusion (up to Week 32)
Population: FAS
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
participants
  All responders | 24 | 22
  Responders, CR | 10 | 15
  Responders, nPR | 1 | 1
  Responders, PR | 13 | 6
  All Non-responders | 7 | 8
  Non-responders, SD | 3 | 2
  Non-responders, PD | 2 | 5
  Non-responders, NE | 2 | 1

12. Secondary Outcome: Number of Participants Classified as Responders Having CR Who Tested Negative for Minimal Residual Disease (MRD)
Description: MRD refers to small number of leukemic cells that remain in the participant during treatment or after treatment when the participant has achieved CR. For all participants who achieved CR, the follow-up bone marrow sample was tested for malignant B cells (CD5+CD19+) to determine if there was any MRD.
Time Frame: From start of treatment (Day 1 of Week 0) until 3 months after start of last infusion (up to course 6 or Week 32)
Population: FAS. Only participants with CR at Visit 34 were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 10 | 15
participants | 2 | 6

13. Secondary Outcome: Ctrough and Cmax at the First Infusion (Visit 2, Week 0) and Sixth Infusion (Visit 29, Week 20)
Description: Cmax is defined as the maximum concentration of drug in plasma samples. Ctrough is defined as the trough plasma concentration (measured concentration at the end of a dosing interval [taken directly before next administration]). No drug is present before the first infusion; therefore, there are no Ctrough results for the first infusion.
Time Frame: Visit 2 (Week 0; up to 4 weeks after dose) and Visit 29 (Week 20; up to 9 months after dose)
Population: as for outcome 5
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams per liter (mg/L)
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 29
Milligrams per liter (mg/L)
  First infusion, Cmax, n=31, 29 | 67.5 (0.47) | 57.2 (0.47)
  Sixth infusion, Cmax, n=22, 19 | 201 (0.30) | 427 (0.34)
  Sixth infusion, Ctrough, n=22, 19 | 19.9 (12.69) | 62.2 (10.36)

14. Secondary Outcome: AUC(0-inf) and AUC(0-672) After the First Infusion (Visit 2, Week 0) and Sixth Infusion (Visit 29, Week 20)
Description: AUC is defined as the area under the ofatumumab concentration-time curve as a measure of drug exposure. AUC(0-672) is AUC from start of infusion to 672 hours after start of infusion; AUC(0-inf) is AUC from start of infusion extrapolated to infinity.
Time Frame: Visit 2 (Week 0; up to 4 weeks after dose) and Visit 29 (Week 20; up to 9 months after dose)
Population: FAS. Data were provided for the number of participants attending each visit for whom the parameter could be calculated. Participants withdrawn during the study were not analyzed.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milligrams * hour per liter (mg.h/L)
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 24 | 26
Milligrams * hour per liter (mg.h/L)
  First infusion, AUC(0-inf), n=24, 26 | 2453 (1.28) | 1915 (0.74)
  First infusion, AUC(0-672), n=24, 26 | 2452 (1.28) | 1915 (0.74)
  Sixth infusion, AUC(0-inf), n=16, 16 | 145236 (0.54) | 397577 (0.35)
  Sixth infusion, AUC(0-672), n=20, 19 | 74728 (0.39) | 149019 (0.75)

15. Secondary Outcome: t1/2 After the First Infusion (Visit 2, Week 0) and Sixth Infusion (Visit 29, Week 20)
Description: t1/2 is defined as terminal half-life and is the time required for the amount of drug in the body to decrease by half.
Time Frame: Visit 2 (Week 0; up to 4 weeks after dose) and Visit 29 (Week 20; up to 9 months after dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 24 | 26
hours
  First infusion, t1/2, n=24, 26 | 19.4 (1.13) | 18.8 (0.62)
  Sixth infusion, t1/2, n=16, 16 | 551 (0.31) | 746 (0.30)

16. Secondary Outcome: CL After the First Infusion (Visit 2, Week 0) and Sixth Infusion (Visit 29, Week 20)
Description: CL is the clearance of drug from plasma, which is defined as the volume of plasma from which the drug is cleared per unit time.
Time Frame: Visit 2 (Week 0; up to 4 weeks after dose) and Visit 29 (Week 20; up to 9 months after dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Milliliters per hour (mL/h)
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 24 | 26
Milliliters per hour (mL/h)
  First infusion, CL, n=24, 26 | 122 (1.28) | 157 (0.74)
  Sixth infusion, CL, n=20, 19 | 6.7 (0.39) | 6.7 (0.75)

17. Secondary Outcome: Vss After the First Infusion (Visit 2, Week 0) and Sixth Infusion (Visit 29, Week 20)
Description: Vss is defined as the volume of distribution at steady state of ofatumumab.
Time Frame: Visit 2 (Week 0; up to 4 weeks after dose) and Visit 29 (Week 20; up to 9 months after dose)
Population: as for outcome 14
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 24 | 26
liters
  First infusion, Vss, n=24, 26 | 3.88 (0.37) | 4.57 (0.30)
  Sixth infusion, Vss, n=16, 16 | 5.15 (0.27) | 5.77 (0.38)

18. Secondary Outcome: Number of Participants With Progression or Death
Description: Disease progression is characterized by at least one of the following, per the Guidelines for the Diagnosis and Treatment of Chronic Lymphocytic Leukemia: a >=50% increase in the sum of the products of at least two lymph nodes on two consecutive determinations 2 weeks apart (at least one node must be >=2 centimeters); or the appearance of new palpable lymph nodes; or a >=50% increase in liver and/or spleen size (measurement below the costal margin); or the appearance of palpable hepatomegaly or splenomegaly not previously present; or a >=50% increase in the numbers of circulating lymphocytes to at least 5.0 * 10^9/Liter; or transformation to a more aggressive histology (e.g., Richter's syndrome or prolymphocytic leukemia with >55% prolymphocytes). For participants who were lost to follow-up, PFS was censored at the date of the last attended visit at which the endpoint was assessed. The Kaplan-Meier method was used to estimate PFS.
Time Frame: as for outcome 3
Population: FAS
Measure: Number; unit: Participants
Arm/Group | Ofatumumab 500 mg + FC | Ofatumumab 1000 mg + FC
Number analyzed (Participants) | 31 | 30
Participants | 3 | 7

ADVERSE EVENTS:
Description: During the Extended Follow-up Phase, from 2 years to 5 years after first treatment, only serious adverse events (SAEs) were collected; no non-serious AEs were collected during this period.
Groups:
- Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC): Ofatumumab intravenous (iv) infusion initiated at 300 milligrams (mg) for course 1, followed by dose of 500 mg for courses 2-6 in combination with fludarabine iv (25 mg/meters squared [m^2] daily on Days 1-3) and cyclophosphamide iv (250 mg/m^2 daily on Days 1-3) administered every 4 weeks for a total of 6 courses
- Ofatumumab 500 mg + FC: Extended Follow-up Phase: Participants were monitored in the Extended Follow-up Phase every 6 months for survival until alternative Chronic Lymphocyte Leukemia (CLL) therapy was initiated, or until Month 60.
- Ofatumumab 1000 mg + FC: Extended Follow-up Phase: Participants were monitored in the Extended Follow-up Phase every 6 months for survival until alternative CLL therapy was initiated, or until Month 60.
Arm/Group | Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC) | Ofatumumab 1000 mg + FC | Ofatumumab 500 mg + FC: Extended Follow-up Phase | Ofatumumab 1000 mg + FC: Extended Follow-up Phase
Serious Adverse Events (participants affected / at risk) | 17/31 | 23/30 | 7/31 | 5/30
Other Adverse Events (participants affected / at risk) | 31/31 | 30/30 | 0/0 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC) (N=31) | Ofatumumab 1000 mg + FC (N=30) | Ofatumumab 500 mg + FC: Extended Follow-up Phase (N=31) | Ofatumumab 1000 mg + FC: Extended Follow-up Phase (N=30)
Neutropenia (Blood and lymphatic system disorders) | 10 | 16 | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 3 | 7 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 4 | 3 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 3 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 2 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 1
Anaemia haemolytic autoimmune (Blood and lymphatic system disorders) | 1 | 0 | 1 | 0
Sepsis (Infections and infestations) | 0 | 2 | 0 | 0
Herpes virus infection (Infections and infestations) | 0 | 1 | 0 | 0
Infection (Infections and infestations) | 0 | 1 | 0 | 0
Bronchitis acute (Infections and infestations) | 0 | 1 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 1
Pneumonia fungal (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 0
Acarodermatitis (Infections and infestations) | 1 | 0 | 0 | 0
Eczema infected (Infections and infestations) | 1 | 0 | 0 | 0
Gastroenteritis rotavirus (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0
Pyrexia (General disorders) | 3 | 0 | 0 | 0
Disease progression (General disorders) | 0 | 1 | 0 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0 | 0
Arthritis reactive (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Renal cell carcinoma stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 1 | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 0 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Alcohol abuse (Psychiatric disorders) | 0 | 1 | 0 | 0
Subclavian vein thrombosis (Vascular disorders) | 1 | 0 | 0 | 0
Acute myeloid leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0
Progressive multifocal leukoencephalopathy (Infections and infestations) | 0 | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Exostosis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 500 mg + Fludarabine and Cyclophosphamide (FC) (N=31) | Ofatumumab 1000 mg + FC (N=30) | Ofatumumab 500 mg + FC: Extended Follow-up Phase (N=0) | Ofatumumab 1000 mg + FC: Extended Follow-up Phase (N=0)
Neutropenia (Blood and lymphatic system disorders) | 14 | 23 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 8 | 16 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 12 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 5 | 5 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 5 | 5 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 4 | 5 | 0 | 0
Nausea (Gastrointestinal disorders) | 14 | 13 | 0 | 0
Vomiting (Gastrointestinal disorders) | 9 | 6 | 0 | 0
Constipation (Gastrointestinal disorders) | 5 | 5 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 0 | 0
Dispepsia (Gastrointestinal disorders) | 4 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 2 | 0 | 0
Pyrexia (General disorders) | 9 | 7 | 0 | 0
Fatigue (General disorders) | 8 | 6 | 0 | 0
Chills (General disorders) | 4 | 5 | 0 | 0
Oedema (General disorders) | 3 | 2 | 0 | 0
Oedema peripheral (General disorders) | 4 | 1 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 10 | 8 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 6 | 3 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 0 | 0
Nasopharyngitis (Infections and infestations) | 5 | 4 | 0 | 0
Bronchitis (Infections and infestations) | 4 | 2 | 0 | 0
Sinusitis (Infections and infestations) | 4 | 2 | 0 | 0
Upper respiratory tract infections (Infections and infestations) | 4 | 2 | 0 | 0
Herpes zoster (Infections and infestations) | 4 | 1 | 0 | 0
Rhinitis (Infections and infestations) | 3 | 2 | 0 | 0
Pneumonia (Infections and infestations) | 2 | 2 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 4 | 0 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 5 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0 | 0
Headache (Nervous system disorders) | 7 | 5 | 0 | 0
Blood creatinine increased (Investigations) | 1 | 4 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 2 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 4 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.